CLINICAL TRIAL: NCT02337114
Title: REACT - Recovery Enhancement From TBI Using ACT. A Pilot Study.
Brief Title: Recovery Enhancement From Traumatic Brain Injury Using Acceptance and Commitment Therapy - a Pilot Study.
Acronym: REACT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Brain Injury Rehabilitation Trust (Other)
Responsible Party: Principal Investigator, Hamish J McLeod PhD CPsychol, Programme Director for Doctorate in Clinical Psychology and Senior Lecturer, University of Glasgow
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/WS/1152
Record Dates: First submitted 2014-12-12; First posted 2015-01-13 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Brain Injuries, Traumatic
Keywords: Acceptance and Commitment Therapy
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Acceptance and Commitment Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Treatment as Usual and Acceptance & Commitment Therapy
  Interventions: Behavioral: Acceptance and Commitment Therapy; Behavioral: Treatment as Usual
- Comparison group (Other): Treatment as Usual
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — A psychotherapeutic intervention that aims to enhance individuals' willingness to have difficult experiences but persist with behaviours that reflect what is important to them.
  Arms: Intervention group
Behavioral: Treatment as Usual — A client-centred goal planning system linked to community reintegration and based on a holistic rehabilitation model including counselling, medical management, cognitive behavioural therapy and pharmacotherapy.

SUMMARY:
Is Acceptance and Commitment Therapy (ACT) feasible and acceptable for adults with severe Traumatic Brain Injury (sTBI) in inpatient services? sTBI is associated with depression, anxiety and low self awareness. A key factor in recovery is adjustment to the effects of injury. Psychological intervention may facilitate this change; however what works is unclear. ACT seeks to improve psychological flexibility; the ability to be present with difficult thoughts and emotions, rather than fighting them, and to accept ourselves as we are, not what we believe we should be. Current research is limited, but what is published suggests it may be useful for this group.

Due to the limited research this pilot study aims to conduct preliminary analysis on the acceptability and feasibility of ACT for people with sTBI whilst also examining the suitability of the study protocol in order to make recommendations for future studies. Clients and staff from three Brain Injury Rehabilitation Trust (BIRT) centres will be recruited, one of which will serve as the intervention centre.

Clients in the intervention group will be asked to complete questionnaires a week before and after participation in the 6 week ACT programme. Clients in the comparison group will be asked to complete questionnaires a week before and after receiving 6 weeks of treatment as usual (TAU). The treatment group will also receive TAU. All participants will be invited to participate in a focus group at the end of this 8 week period to discuss their involvement in the study.

Staff will be asked to complete a parallel version of one of the client questionnaires within a similar timeframe. In addition staff at the intervention centre will be invited to attend a focus group and complete an additional questionnaire after the eight week period.

DETAILED DESCRIPTION:
A pilot study design will initially assess the feasibility and acceptability of the ACT and study protocol with this client group in order to inform a future clinical trial.

The methodology involves both quantitative and qualitative methods and will involve inpatients at Brain Injury Rehabilitation Trust (BIRT) units, staff involved in the day to day care of inpatients and clinicians involved in the administration of therapy. Quantitative methods (questionnaires) were chosen to assess any possible change in assessment measures. The measures chosen have been previously used. They have good validity (the ability to answer the questions asked) and reliability, and therefore are practically suitable for measuring outcomes of therapy. Qualitative methods (focus groups) were also chosen, owing to the pilot nature of this research, in order to obtain personal opinion on the acceptability of the intervention and the treatment protocol, from those participating.

The intervention will be administered, alongside TAU, to inpatients at a BIRT centre in Glasgow and will be compared to a comparison group which will receive TAU only (who will be based in BIRT centres in either York and/or Leeds). The rational for choosing a BIRT centre in Glasgow for the intervention group is one of convenience as all researchers involved in the study are based in Glasgow. This will help facilitate data collection and reduce cost. Given that all BIRT centres adhere to a similar philosophy of care and rehabilitation and service user profiles are relatively similar, it was believed that recruiting elsewhere for the purpose of comparison would be appropriate. Recruiting treatment and comparison groups from separate centres also ensures that clients receiving TAU only do not learn ACT strategies accidentally through discussion with peers or staff. If this were to happen any indication of change could not be attributed to the difference in treatments provided.

Five participant groups will be recruited:

* clients in the inpatient setting (treatment group),
* clients in the inpatient setting (comparison group),
* care staff working directly with clients (treatment group),
* care staff working directly with clients (comparison group)
* psychology staff involved in administering the intervention.

All participants will be provided with an information sheet and consent will be sought prior to their participation in the study. All interventions, assessments and focus groups will be completed at the participants respective centres. All recruitment, with the exception of the psychology staff who are a convenient sample, will be conducted by a staff member not involved in the direct write up of the study. Further to this all outcome measures and focus groups will be conducted by researchers not involved in the provision of treatment.

Psychology staff at the intervention centre who have completed training on ACT will be further informed of the study. If they choose to participate they will recruit clients at BIRT in Glasgow, completing a record form identifying inclusion and exclusion criteria met. This form will allow the staff to outline any barriers or difficulties encountered as part of this process. Information sheets will then be provided to recruited clients, in addition to care staff who work with them.

The study will also be explained to heads of service at each of the comparison sites, providing them both with an integrated protocol. They will identify a point of contact who will complete recruitment as detailed above.

Each participant will be given between 24hours and 1 week to decide whether to participate.

Researchers will first meet with care staff informed of the study at each centre to discuss their own consent and provide consent form to them. At this point only risk information for each client will be discussed with the care staff with the purpose of ensuring the safety of both the clients and researchers at first point of contact.

Researchers will meet with recruited clients individually to discuss consent and complete questionnaires.

Researchers will again meet with care staff to discuss client demographic information and to complete one questionnaire, if clients have consented for this to take place.

The trained psychology staff will provide 6 weeks of ACT training to clients in the treatment group weekly. Each group will have up to 4 clients per group.

Researchers will meet with both groups after this time period to repeat testing of the questionnaires with both staff.

Details concerning what treatments, aside from ACT, were provided to each client during the 6 week period will be collected from case files and through discussion with staff.

Clients at all centres will be invited to take part in a focus group at this time to discuss their participation in the study.

Care staff at the intervention centre will be invited to participate in a focus group.

Psychology staff at the intervention centre will be invited to participate in a focus group and complete a questionnaire.

Further research tasks to be completed by staff:

Any observations as part of applying the study protocol will also be documented. For example, the participant flow, drop out rates, the administration of questionnaires, the storage of materials and ethical issues will all be commented upon as per the objective of the overall pilot study.

Guidelines for reporting Serious Adverse Events (SAEs) will be piloted as part of this study. In order to establish base rates for this group, a record will be kept of any SAE experience by participants of intervention or comparison group. A checklist of potential SAEs will be used at both times of testing for treatment and control group in order to establish whether any SAEs occurred.

ELIGIBILITY:
Inclusion Criteria:

All clients must:

* have sustained a severe TBI after the age of 18; indicated by presence of posttraumatic amnesia for a day or more OR loss of consciousness for 30 minutes or more following injury OR scores of eight or less on the Glasgow Coma Scale.
* have sufficient English language skills to enable valid participation using standard tests and questionnaires
* be admitted to BIRT for neuropsychological rehabilitation
* have sufficient cognitive capacity to complete questionnaires independently and participate in discussions as part of the ACT intervention.

All psychology staff must have:

* completed 1.5 day ACT training
* time and resources to:
* administer ACT intervention to at least one group of 3-4 clients once a week for a six week period within the time frame suggested for this pilot study
* participate in a focus group following intervention providing their views of the study protocol
* complete the SAFE questionnaire identifying barriers to treatment implementation

Care staff not involved in delivering the intervention (including nursing staff and rehabilitation support workers)

* will have the time and resources to complete 2 questionnaires
* work directly with the clients receiving the intervention
* have commenced at BIRT employment prior to the first intervention session.
* will have the time and resources to participate in the focus group, if based at Graham Anderson House

Exclusion Criteria:

Clients will be excluded from the study if they:

* lack capacity to consent to participate in research as assessed by staff at BIRT or by the researcher when discussing consent with the participant
* will remain in the unit for less than eight weeks
* have challenging behaviour that may put the researcher or participant at risk or prevent participation in the study.

Psychology staff will be excluded if:

* they have not received the appropriate training
* they consider that do not have the time and resources to partake in all the research tasks.

Care staff will be excluded from this study if:

* they have commenced employment after the study procedures have commenced
* they believe they do not have the time and resources to complete research tasks
* they do not work directly with clients participating in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Acceptability of ACT as measured by focus-group discussions with clients and staff; number of participants withdrawing from study | 9 weeks
  Qualitative thematic analysis of focus-group discussions with clients and staff; number of participants withdrawing from study
Suitability of ACT as measured by Acceptance and Action Questionnaire - Acquired Brain Injury | 9 weeks
  Quantitative comparison between groups of results of Acceptance and Action Questionnaire - Acquired Brain Injury
Feasibility of ACT as measured by focus-group discussions with clients and staff; number of participants considering intervention satisfactory/appropriate | 9 weeks
  Qualitative thematic analysis of focus-group discussions with clients and staff; number of participants considering intervention satisfactory/appropriate

SECONDARY OUTCOMES:
Suitability of ACT, as measured by Hospital Anxiety and Depression Scale | 9 weeks
  Quantitative comparison between groups of results of the Hospital Anxiety and Depression Scale
Suitability of ACT as measured by the Motivation for Traumatic Brain Injury Rehabilitation Questionnaire | 9 weeks
  Quantitative comparison between groups of results of Motivation for Traumatic Brain Injury Rehabilitation Questionnaire
Suitability of ACT as measured by Awareness Questionnaire | 9 weeks
  Quantitative comparison between groups of results of Awareness Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hamish McLeod, PhD CPsychol, Principal Investigator — University of Glasgow
Locations (1):
- Brain Injury Rehabilitation Trust, Glasgow, United Kingdom